CLINICAL TRIAL: NCT00036062
Title: A Phase II Study to Determine the Efficacy and Safety of Sivelestat in Subjects With Acute Lung Injury
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6025; H6W-MC-MCAA
Record Dates: First submitted 2002-05-07; First posted 2002-05-08 (Estimated); Last update posted 2006-07-19 (Estimated); Status verified 2006-07

CONDITIONS: Respiratory Distress Syndrome, Adult; Acute Lung Injury
Keywords: Sivelestat; acute lung injury
MeSH Terms: conditions — Respiratory Distress Syndrome; Acute Lung Injury | interventions — sivelestat

INTERVENTIONS:
Drug: Sivelestat

SUMMARY:
The purpose of this study is to determine whether sivelestat will reduce the amount of time a patient must spend on a ventilator and/or increase the chance of survival of patients with acute lung injury.

DETAILED DESCRIPTION:
Acute lung injury often develops as a result of severe infection, sepsis, severe injuries, inhalation of foreign substances into the lungs, or pneumonia. The tissues and blood vessels in the lungs become inflamed, and the body does not receive enough oxygen. Patients with this condition are placed on a ventilator to assist with breathing.

Patients entered into this study will be randomly assigned to one of two treatment groups: a sivelestat group or a placebo group. Once entered into the study, patients are monitored for up to 6 months.

ELIGIBILITY:
Inclusion Criteria

* show evidence of acute lung injury
* be on mechanical ventilation

Exclusion Criteria

* have undergone certain organ transplants
* have severe underlying medical problems
* be unlikely to survive
* be pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600
Dates: Start 2001-08; Study Completion 2002-12

CONTACTS AND LOCATIONS:
Locations (110):
- United States (65):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Tucson, Arizona
  - Orange, California
  - Sacramento, California
  - San Diego, California
  - Denver, Colorado
  - Englewood, Colorado
  - New Haven, Connecticut
  - Washington D.C., District of Columbia
  - Bay Pines, Florida
  - Clearwater, Florida
  - Fort Lauderdale, Florida
  - Augusta, Georgia
  - Austell, Georgia
  - Chicago, Illinois
  - Elk Grove Village, Illinois
  - Maywood, Illinois
  - North Chicago, Illinois
  - Indianapolis, Indiana
  - Des Moines, Iowa
  - Kansas City, Kansas
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Baton Rouge, Louisiana
  - Lake Charles, Louisiana
  - Shreveport, Louisiana
  - Portland, Maine
  - Baltimore, Maryland
  - Silver Spring, Maryland
  - Towson, Maryland
  - Boston, Massachusetts
  - Detroit, Michigan
  - Kalamazoo, Michigan
  - St Louis, Missouri
  - Camden, New Jersey
  - Hackensack, New Jersey
  - Holmdel, New Jersey
  - Buffalo, New York
  - Elmhurst, New York
  - Manhasset, New York
  - Mineola, New York
  - New York, New York
  - Rochester, New York
  - The Bronx, New York
  - Greensboro, North Carolina
  - Winston-Salem, North Carolina
  - Akron, Ohio
  - Cincinnati, Ohio
  - Toledo, Ohio
  - Portland, Oregon
  - Allentown, Pennsylvania
  - Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Providence, Rhode Island
  - Sioux Falls, South Dakota
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Houston, Texas
  - Irving, Texas
  - Lubbock, Texas
  - San Antonio, Texas
  - Newport News, Virginia
  - Morgantown, West Virginia
- Australia (15):
  - Garran, Australian Capital Territory
  - Camperdown, New South Wales
  - Kingswood, New South Wales
  - Kogarah, New South Wales
  - St Leonards, New South Wales
  - Wentworthville, New South Wales
  - Southport, Queensland
  - Adelaide, South Australia
  - Bedford Park, South Australia
  - Woodville, South Australia
  - Heidelberg, Victoria
  - Parkville, Victoria
  - Prahran, Victoria
  - Fremantle, Western Australia
  - Perth, Western Australia
- Belgium (8):
  - Aaist
  - Antwerp
  - Arion
  - Braine-l'Alleud
  - Bruges
  - Brussels
  - Ghent
  - Liège
- Canada (9):
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Winnipeg, Manitoba
  - Halifax, Nova Scotia
  - Hamilton, Ontario
  - Toronto, Ontario
  - Windsor, Ontario
  - Montreal, Quebec
  - Sherbrooke, Quebec
- New Zealand (4):
  - Christchurch, Canterbury
  - Auckland
  - Hastings
  - Wellington
- Spain (9):
  - Badajoz, Badajoz
  - Manresa, Barcelona
  - Sabadell, Barcelona
  - Getafe, Madrid
  - Madrid, Madrid
  - El Palmar, Murcia
  - Murcia, Murcia
  - Palma de Mallorca, Palma de Mallorca
  - Barcelona